CLINICAL TRIAL: NCT03524755
Title: Effects of a Progressive Resistance Training in Cachectic Cancer Patients During Radiotherapy - a Randomized Controlled Pilot Trial
Brief Title: Physical Exercise for Patients Who Suffer From Weight Loss Due to Head and Neck Cancer Undergoing Medical Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Dr. med. Dipl.-Phys. Maximilian Niyazi, PD Dr. med. Dipl. Phys. Karim- Maximilian Niyazi, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cancer Cachexia Exercise
Record Dates: First submitted 2018-04-29; First posted 2018-05-15 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Head and Neck Cancer; Cachexia; Cancer; Resistance Training
MeSH Terms: conditions — Head and Neck Neoplasms; Cachexia; Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): Warm up period for 5 minutes on a bicycle ergometer or an upper body cycle with individual selectable wattage. A leg press, a latissimus pull-down and a chest press formed the three equipment supported core exercises. All exercises were performed with 8-12 repetitions and 3 sets. 3 training sessions (30min for each session) per week for during the course of radiotherapy (~6 weeks).
  Interventions: Other: Exercise
- Control Group (No Intervention): The control group received usual care.

INTERVENTIONS:
Other: Exercise
  Arms: Training Group

SUMMARY:
Cancer cachexia is a prevalent symptom of head and neck neoplasms. The reduction in skeletal muscle mass is one of the main characteristics which can lead to poor physical functioning. The purpose of this study was to determine the feasibility of progressive resistance training in cachectic head and neck cancer patients during radiotherapy in a pilot randomized controlled design.

Baseline data for all participants were ascertained via medical records and patient interview. This included demographic information, Union internationale contre le cancer-status (UICC-status), comorbidities and the results of blood samples. Outcomes were measured at admission. One study coordinator completed all assessments to enhance patient compliance. Body weight loss percentage was calculated via the individuals' body weight 6 months before (in retrospect) and the current body weight. Participants completed two questionnaires: The Multidimensional Fatigue Inventory and the Functional Assessment of Anorexia/Cachexia Therapy questionnaire. Six-Minute Walk Test was applied. To document changes in muscle force, strength of the functional muscle group for elbow flexion in supine position as well as of knee extension in sitting position (in each case right and left) was tested via hand-held dynamometry for isometric maximal muscle strength. Bioelectrical impedance analysis was executed to assess the adaption in body composition.

The exercise intervention was undertaken in the hospitals department of physical and rehabilitation medicine and based on standardized but individualized training protocols. It consisted of a warm up period for 5 minutes on a bicycle ergometer or an upper body cycle with individual selectable wattage. A leg press, a latissimus pull-down and a chest press formed the three equipment supported core exercises. All exercises were performed with 8-12 repetitions and 3 sets.

ELIGIBILITY:
Inclusion Criteria:

* planned inpatient or outpatient radiotherapy
* ≥ 18 years of age
* diagnosed state of cachexia (weight loss greater than 5 % over the past 6 months) or pre-cachexia (unintentional weight loss of 5 % or less of usual body weight during the last 6 months)

Exclusion Criteria:

* metastatic disease
* severe neurological problems or other contraindications for resistance training

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07-10 (Actual); Primary Completion 2015-05-07 (Actual); Study Completion 2015-05-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Cancer-related fatigue at post-radiotherapy and follow-up | Baseline, post-radiotherapy (~6weeks), follow-up (~8 weeks)
  The Multidimensional Fatigue Inventory (MFI) which consists of 20 items that measure subgroups (general, physical and mental fatigue as well as reduced motivation and reduced activity) of fatigue with a 5-point Likert scale.

SECONDARY OUTCOMES:
Change from Baseline Anorexia/Cachexia at post-radiotherapy and follow-up | Baseline, post-radiotherapy (~6weeks), follow-up (~8 weeks)
  Functional Assessment of Anorexia/Cachexia Therapy (FAACT) questionnaire which registers well-being for physical, social/family, emotional and functional aspects of quality of life and additional concerns in cachexia with 5-point Likert scale for 39 items

CONTACTS AND LOCATIONS:
Overall Officials: Claus Belka, Prof. Dr., Principal Investigator — Klinikum der Universität München, Klinik und Poliklinik für Strahlentherapie und Radioonkologie

IPD SHARING:
Plan to Share IPD: No
My institution does not require data sharing and because of ethical concerns.

REFERENCES:
- [Background] Couch M, Lai V, Cannon T, Guttridge D, Zanation A, George J, Hayes DN, Zeisel S, Shores C. Cancer cachexia syndrome in head and neck cancer patients: part I. Diagnosis, impact on quality of life and survival, and treatment. Head Neck. 2007 Apr;29(4):401-11. doi: 10.1002/hed.20447. PMID 17285641
- [Background] Speck RM, Courneya KS, Masse LC, Duval S, Schmitz KH. An update of controlled physical activity trials in cancer survivors: a systematic review and meta-analysis. J Cancer Surviv. 2010 Jun;4(2):87-100. doi: 10.1007/s11764-009-0110-5. Epub 2010 Jan 6. PMID 20052559
- [Background] Smets EM, Garssen B, Cull A, de Haes JC. Application of the multidimensional fatigue inventory (MFI-20) in cancer patients receiving radiotherapy. Br J Cancer. 1996 Jan;73(2):241-5. doi: 10.1038/bjc.1996.42. PMID 8546913
- [Background] Ribaudo JM, Cella D, Hahn EA, Lloyd SR, Tchekmedyian NS, Von Roenn J, Leslie WT. Re-validation and shortening of the Functional Assessment of Anorexia/Cachexia Therapy (FAACT) questionnaire. Qual Life Res. 2000;9(10):1137-46. doi: 10.1023/a:1016670403148. PMID 11401046
- [Background] Schmidt K, Vogt L, Thiel C, Jager E, Banzer W. Validity of the six-minute walk test in cancer patients. Int J Sports Med. 2013 Jul;34(7):631-6. doi: 10.1055/s-0032-1323746. Epub 2013 Feb 26. PMID 23444095
- [Derived] Grote M, Maihofer C, Weigl M, Davies-Knorr P, Belka C. Progressive resistance training in cachectic head and neck cancer patients undergoing radiotherapy: a randomized controlled pilot feasibility trial. Radiat Oncol. 2018 Nov 6;13(1):215. doi: 10.1186/s13014-018-1157-0. PMID 30400971